CLINICAL TRIAL: NCT05276895
Title: Evaluation of the Efficacy of Natural Senolytic Agents and NLRP3 Inhibitors in Treatment of Osteoarthritis: Randomized, Double Blinded ,Placebo Controlled Trial
Brief Title: Effect of Natural Senolytic Agents & NLRP3 Inhibitors on Osteoarthritis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailability of drugs
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Adel A.Gomaa, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17101628
Record Dates: First submitted 2022-01-11; First posted 2022-03-14 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis
Keywords: Intervention, natural senolytics, NLRP3 inhibitors, trial
MeSH Terms: conditions — Osteoarthritis | interventions — Quercetin; fisetin; Glycyrrhizic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (Quercetin +Fisetin) (Active Comparator): 20 participants with symptomatic knee osteoarthritis and ultrasonography defined effusion-synovitis will take natural Senolytic agents.
  The senolytic agents act by Hit-and-run strategy therefore, intermittent dosing regimens will be applied. 1250 mg/day quercetin + 1000mg/day Fisetin for 3 consecutive days every 3 weeks.over 12 weeks
  Interventions: Dietary Supplement: Quercetin and Fisetin tab.
- Quercetin +Fisetin +Glycyrrhizin) (Active Comparator): 20 participants with symptomatic knee osteoarthritis and ultrasonography-defined effusion-synovitis will take Quercetin 1250 mg + Fisetin 1000 mg for 3 consecutive days followed by 100mg/day Glycyrrhizin for one week every 3 weeks over 12 weeks .
  Interventions: Dietary Supplement: Quercetin Cap/Tab,Fisetin Cap/tab and Glycyrrhizin capsules
- Placebo (Placebo Comparator): Placebo controlled group
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin and Fisetin tab. — 1250 mg/day quercetin + 1000mg/day Fisetin for 3 consecutive days every 3 weeks over 15 weeks .
  Arms: (Quercetin +Fisetin)
Dietary Supplement: Quercetin Cap/Tab,Fisetin Cap/tab and Glycyrrhizin capsules — quercetin + Fisetin for 3 consecutive days followed by 100mg/day glycyrrhizin for one week every 3 weeks over 15 weeks
  Arms: Quercetin +Fisetin +Glycyrrhizin)
Other: Placebo — Placebo capsule for one week every 3 weeks over 15 weeks
  Arms: Placebo

SUMMARY:
Objective: To determine the efficacy of natural senolytic agents and NLRP3 Inflammasome inhibitors for reducing knee symptoms and effusion-synovitis in patients with symptomatic knee osteoarthritis and knee effusion-synovitis.

Design: Randomized, double-blind, placebo-controlled trial. Setting: Single-center study with outpatients from university hospital , Faculty of Medicine , Assiut, Egypt .

Participants: 60 participants with symptomatic knee osteoarthritis and ultrasonography-defined effusion-synovitis. Randomized to 3 arms ( natural Senolytic agents alone, natural senolytic plus natural NLRP3 Inflammasome inhibitors and placebo) Intervention: The senolytic agents act by Hit-and-run strategy therefore, intermittent dosing regimens will be applied. 1250 mg/day quercetin + 1000mg/day Fisetin for 3 consecutive days every 3 weeks (n = 20), quercetin + Fisetin for 3 consecutive days followed by 100mg/day glycyrrhizin for one week every 3 weeks (n=20) or matched placebo (n = 20) over 15 weeks Measurements: . The primary outcome measures were change in knee pain (assessed by visual analogue scale VAS) and effusion-synovitis volume on magnetic resonance imaging (MRI). Secondary outcomes are listed as follows: knee pain, function, and stiffness assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), OARSI-OMERACT (Outcome Measures in Rheumatology Clinical trials- Osteoarthritis Research Society International) responders to treatment, cartilage compositional change assessed by cartilage T2 relaxation time (ms), pain medication usage, change in quality of life (Assessment of Quality of Life (AQoL-4D) questionnaire),

DETAILED DESCRIPTION:
Osteoarthritis is a progressive degenerative disease of the joint leading to cartilage damage, pain and loss of function affecting an estimated 250 million people worldwide and 27 million people in the United States .Currently, there are no effective FDA-approved therapies that are disease-modifying interventions to block the joint destruction pathway because of osteoarthritis. The most prevalent first-line treatment for OA is to mitigate pain and restore function with a combination of weight management, physical therapy, mind-body exercises, and analgesia with paracetamol or NSAIDs (topical or oral) . Another prominent treatment strategy is the use of intra-articular corticosteroids (CS) to reduce pain and inflammation via targeting production of interleukins, leukotrienes and prostaglandins.

However, the palliative effects of CS for OA are often short-term, can potentially lead to chondral fissuring and promotion of dose-independent structural changes in cartilage, and there are no consistent reports of efficacy .

One novel potential and appealing approach for treating osteoarthritis is through the local and systemic elimination of senescent cells. Senescent cell burden increases significantly with age and has been shown to promote several age-related pathologies including degenerative joint conditions. Senescent cells are non-proliferative, resistant to apoptosis, and secrete pro-inflammatory factors that promote disease and systemic aging .Cellular senescence can be induced by a variety of extrinsic and intrinsic signals that leads to the production of a collection of various proinflammatory cytokines and other factors that initiate senescence in neighbouring cells and promote disease and tissue dysfunction. Thus, senescent cells and their associate senescence associated secretory phenotype profiles likely play a role in both the clinical manifestation of OA (pain) and disease pathogenesis (tissue dysfunction and cartilage degradation.

The overall safety and efficacy of several senolytic drugs to treat chronic diseases have been demonstrated in several preclinical studies and more recently in phase I-II clinical trials for OA. However, there are no encouraging results with the use of natural senescent agents such as quercetin or fisetin as disease-modifying agents in OA, therefore, our study will investigate the effect of a combination of natural senescent agents and NLRP3 inhibitors on inflammation.

Inflammasomes play a crucial role in innate immunity by serving as signalling platforms which deal with a plethora of pathogenic products and cellular products associated with stress and damage. By far, the best studied and most characterized inflammasome is NLRP3 inflammasome, which consists of NLRP3 (nucleotide-binding domain leucine-rich repeat (NLR) and pyrin domain containing receptor 3). The hyperactivation of NLRP3 inflammasome is involved in a wide range of inflammatory diseases. The search and development of anti-inflammatory drugs from natural sources of plants has received extensive attention. licorice extract has high activity and wide therapeutic effects.it has reported that glycyrrhizin could ameliorate fibrosis and inflammation via inhibiting NLRP3 inflammasome activation and NF-κB signalling pathway.

our aim is to determine the efficacy of Natural senolytic agents and NLRP3 Inflammasome inhibitors for reducing knee symptoms and effusion- synovitis in patients with symptomatic knee Osteoarthritis and knee effusion /synovitis.

ELIGIBILITY:
Inclusion Criteria:

* male or female, ages 40-80;
* Are willing to comply with all study related procedures and assessments;
* ambulatory as defined by ability to complete functional performance testing;
* Radiographic evidence of Kellgren-Lawrence grade II-IV osteoarthritis in one or both knees;
* Scores 4-10 on the Numerical Rating Scale (NRS) for pain;

Exclusion Criteria:

* Pregnant or nursing females.
* Subjects who do not have the capacity to consent themselves.
* Subjects who are unable to tolerate oral medication.
* Subjects with uncontrolled medical conditions .
* Surgery on the Study Knee in the past 6 months.
* intra-articular injection of corticosteroids or hyaluronic acid in the past 6 months.
* subjects with significant liver or renal disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain on the visual analogu scale at end of treatment | Baseline (at beginning of the trial at day 1),after 3 weeks,after 6 weeks and after 12 weeks(end of the trial)
  Each participant was asked to indicate his or her current level of pain on a100 mm scale.
  0 mm indcates no pain and 100mm indicates the worst pain imaginable.

SECONDARY OUTCOMES:
WOMAC (western Ontario and McMaster Universities Osteoarthritis Index | Will be assessed before (at beginning of the trial at day 1),after 3 weeks,after 6 weeks and after 12 weeks(end of the trial)
  For assessment of knee function, pain,and stiffness.(5 items for pain ,2 items for stiffness and 7 items for functional limitation and when score is higher means more pain and more stiffness and more functional limitation, items like using stairs ,standing from setting, walking, getting in and out of acar ,lying in bed...)
IL-17 | Will be measured before(at beginning of the trial )and at the end of the trial(after 12 weeks)
  Laboratory test (serum sample)

CONTACTS AND LOCATIONS:
Overall Officials: Adel A. Gomaa, Ph.D., Principal Investigator — Assiut University
Locations (1):
- Assiut University, Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will become available to interested investigators upon submitting a reasonable research request by email to A. Gomaa
  (a.gomma@aun.edu.eg).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Dec.2023
Access Criteria: Data will become available to interested investigators upon submitting a reasonable research request by email to A. Gomaa
  (a.gomma@aun.edu.eg).

REFERENCES:
- [Background] Bentley G, Biant LC, Carrington RW, Akmal M, Goldberg A, Williams AM, Skinner JA, Pringle J. A prospective, randomised comparison of autologous chondrocyte implantation versus mosaicplasty for osteochondral defects in the knee. J Bone Joint Surg Br. 2003 Mar;85(2):223-30. doi: 10.1302/0301-620x.85b2.13543. PMID 12678357
- [Background] da Costa BR, Hari R, Juni P. Intra-articular Corticosteroids for Osteoarthritis of the Knee. JAMA. 2016 Dec 27;316(24):2671-2672. doi: 10.1001/jama.2016.17565. PMID 28027351
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Gel'man SI. [The choice of rational modes of artificial pulmonary ventilation in cerebral operations]. Eksp Khir Anesteziol. 1965 Nov-Dec;10(6):57-60. No abstract available. Russian. PMID 5873863
- [Background] Milstein C, Clegg JB, Jarvis JM. C-terminal half of immunoglobulin lambda-chains. Nature. 1967 Apr 15;214(5085):270-2. doi: 10.1038/214270a0. No abstract available. PMID 4166495
- [Background] Stokes J, Drury RA. Gordon Roy Cameron. J Clin Pathol. 1967 Jan;20(1):5-6. doi: 10.1136/jcp.20.1.5. No abstract available. PMID 5334539
- [Background] Niemineva K. [1897--a landmark in Finnish medical literature]. Duodecim. 1966;82(17):823-7. No abstract available. Finnish. PMID 5331226
- [Background] Martinon F, Burns K, Tschopp J. The inflammasome: a molecular platform triggering activation of inflammatory caspases and processing of proIL-beta. Mol Cell. 2002 Aug;10(2):417-26. doi: 10.1016/s1097-2765(02)00599-3. PMID 12191486
- [Background] Panich V, Sungnate T, Na-Nakorn S. Acute intravascular hemolysis and renal failure in a new glucose-6-phosphate dehydrogenase variant: G-6-PD Siriraj. J Med Assoc Thai. 1972 Dec;55(12):726-31. No abstract available. PMID 4650733
- [Background] Winniford MD, Jansen DE, Reynolds GA, Apprill P, Black WH, Hillis LD. Cigarette smoking-induced coronary vasoconstriction in atherosclerotic coronary artery disease and prevention by calcium antagonists and nitroglycerin. Am J Cardiol. 1987 Feb 1;59(4):203-7. doi: 10.1016/0002-9149(87)90785-5. PMID 3101478